CLINICAL TRIAL: NCT03994783
Title: A Multicentre Randomised Controlled Trial to Assess the Efficacy of Adding Rituximab to Standard of Care in Treating Acute Antibody-mediated Rejection in Kidney Transplantation
Brief Title: Transplant Antibody-Mediated Rejection: Guiding Effective Treatments
Acronym: TAR:GET-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped at start of COVID-19 pandemic - non-feasible
Sponsor: Imperial College London (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Kidney Cancer UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-002882-20
Record Dates: First submitted 2019-06-17; First posted 2019-06-21 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplant Rejection; Antibody-mediated Rejection
Keywords: Rituximab; AMR
MeSH Terms: interventions — Rituximab; Methylprednisolone; Immunoglobulins, Intravenous; Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Intravenous Methylprednisolone (500 mg (600 mg/m2 for paediatric participants), n=3) Plasma Exchange (PEX) (60 ml/kg max 4 l (1 - 1.5 plasma volumes for paediatric participants), n=7) Intravenous Immunoglobulin (high dose: 2 g/kg total, or low dose: 100 mg/kg n=7 after each PEX, no dose adjustment for paediatric participants)
  Interventions: Drug: Methylprednisolone; Drug: Intravenous Immunoglobulin; Procedure: Plasma Exchange
- Standard of Care plus Rituximab (SOCR) (Experimental): Intravenous Methylprednisolone (500 mg (600 mg/m2 for paediatric participants), n=3) Plasma Exchange (PEX) (60 ml/kg max 4 l (1 - 1.5 plasma volumes for paediatric participants), n=7) Intravenous Immunoglobulin (high dose: 2 g/kg total, or low dose: 100 mg/kg n=7 after each PEX, no dose adjustment for paediatric participants) Rituximab (375 mg/m2 max 1 g (no dose adjustment for paediatric participants), n=2 14 days +/- 2 days apart)
  Interventions: Drug: Rituximab; Drug: Methylprednisolone; Drug: Intravenous Immunoglobulin; Procedure: Plasma Exchange

INTERVENTIONS:
Drug: Rituximab — 2 intravenous infusions of rituximab or approved biosimilar given 14 days +/- 2 days apart.
  Other Names: Rituximab Biosimilar; Mabthera
  Arms: Standard of Care plus Rituximab (SOCR)
Drug: Methylprednisolone — Intravenous infusion of methylprednisolone
Drug: Intravenous Immunoglobulin — High dose (2 g/kg total) or Low dose (100 mg/kg, n=7)
Procedure: Plasma Exchange — Blood is removed from the patient and filtered to remove the plasma. Red and white blood cells and platelets are returned to the patient with replacement fluid.

SUMMARY:
This trial evaluates the addition of rituximab to standard of care in the treatment of antibody-mediated rejection in kidney transplant patients. The trial will involve adults and children. Half of participants will receive standard of care (methylprednisolone, intravenous immunoglobulin and plasma exchange), while the other half will receive standard of care and rituximab.

DETAILED DESCRIPTION:
Chronic antibody-mediated rejection (cAMR) is the leading cause of kidney transplant failure. Fifty percent of kidney transplant patients who develop acute antibody-mediated rejection (aAMR) will develop evidence of cAMR within 1 year of the acute rejection episode. There is currently no evidence on how to treat aAMR.

The planned research is a randomised controlled trial, which compares an acceptable and commonly used therapy, which will be referred to as "standard of care", with an additional agent, rituximab, added to the "standard of care" treatment. The participants with be randomised in a 1:1 ratio.

"Standard of care" will include optimisation of the participant's baseline anti-rejection medications and therapy to remove the antibodies which have developed against the kidney transplant, which are causing the damage. This is called plasma exchange. The participants will also receive therapy to reduce inflammation and reduce their immune response to their kidney transplant. This will be achieved using corticosteroids and intravenous immunoglobulins, respectively. These therapies have been used to treat aAMR for many decades.

The intervention arm will consist of the "standard of care" treatment, with the addition of a drug called rituximab, which will be administered in 2 separate doses. Rituximab is itself an antibody, which binds to certain cells in the body involved in antibody production, called B cells. Following the administration of rituximab, the number of B cells is reduced, which affects antibody production. Rituximab is commonly used in transplantation for this indication, as well as for other conditions.

Participants in both arms will be followed up to determine if there is a difference in the time to transplant failure and/or transplant function.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent by patient aged 16 years and over; or by a parent or legal guardian for patients who are under 16 years old
* 5 years old or older
* A diagnosis of acute AMR as defined by:
* The presence of ≥1 donor specific antibodies (DSA)
* An adequate renal transplant biopsy with histological features consistent with active AMR with no evidence of chronicity as defined by the Banff histological classification of allograft pathology:
* If C4d positive (2 or 3):
* v score ≥1 and/or
* g score ≥1 and/or
* thrombotic microangiopathy and/or
* ptc score ≥1
* or if co-existent cellular rejection, a g score of ≥1 OR
* If C4d negative (0 or 1):
* microcirculation inflammatory score (g + ptc) ≥2
* or if co-existing cellular rejection, a g score ≥1 and (g + ptc) ≥2 AND
* Chronic glomerulopathy (cg) score 0 or 1a
* Tubulo-interstitial fibrosis <50% and glomerular obsolescence <50%

Exclusion Criteria:

* Patients who have received an ABO incompatible transplant
* Patients who have received rituximab as part of induction or post-transplant for any other indications (e.g. recurrent focal and segmental glomerular sclerosis)
* Patients who have completed PEX treatment prior to the index biopsy on the suspicion of acute AMR in the absence of histology
* Have active infection including bacterial, viral (including CMV (cytomegalovirus) and EBV (Epstein-Barr virus)), fungal or tuberculosis, which in the investigator's opinion could affect the conduct of the trial
* Co-existing BK (BK virus) nephropathy
* Patients with hepatitis B (patients with prior exposure to hepatitis B may be enrolled at the discretion of the PI)
* Have active hepatitis C (patients may be included if a negative hepatitis C recombinant immunoblot assay is confirmed or have a negative hepatitis C virus RNA [qualitative] test)
* Have human immunodeficiency virus (HIV)
* Active malignancy, which would pose a contraindication to any of the trial interventions
* Patients with known allergy, intolerance or contraindication to treatments in the standard of care arm or rituximab as outlined in the Summaries of Product Characteristics (SmPCs)
* Clinically significant comorbidity
* Females must be either post-menopausal for at least 1 year, surgically sterile or, if of child-bearing potential, must not be pregnant or lactating. If sexually active, female participants must agree to use an acceptable method of birth control for 12 months post treatment with rituximab. Female participants must also agree not to breastfeed for 12 months post treatment with rituximab.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Allograft Survival as assessed by statistical model | 4 years
  Statistical model measuring allograft survival as defined as duration from the date of randomisation to the date of eGFR ≤15 mL/min/1.72 m2 (where the eGFR measurement is not due to an acute reversible cause, as determined by the PI, or a follow-up consecutive eGFR measurement of ≤15 mL/min/1.72 m2 is recorded (where the first date is recorded as the date of failure)), or the date of renal replacement therapy (date of starting maintenance dialysis dependency, retransplantation etc), whichever occurs first.

SECONDARY OUTCOMES:
Serum creatinine as assessed by blood test | 1, 3, 6 and 12 months, 2, 3 and 4 years
  Serum creatinine is an allograft function. Change in serum creatinine from baseline at 1, 3, 6 and 12 months post-randomisation and then annually until 4 years
Estimated glomerular filtration rate (eGFR) as assessed by blood test | 1, 3, 6 and 12 months, 2, 3 and 4 years
  eGFR is an allograft function. Change in eGFR from baseline at 1, 3, 6 and 12 months post-randomisation and then annually until 4 years
Proteinuria as assessed by urine test | 1, 3, 6 and 12 months, 2, 3 and 4 years
  Proteinuria is an allograft function. Change in proteinuria from baseline at 1, 3, 6 and 12 months post-randomisation and then annually until 4 years. Proteinuria is a ratio between urinary protein and creatinine.
Change in donor specific antibodies as assessed by blood test | 3 and 12 months
  Change in number of donor specific antibodies from baseline
Change in positivity of donor specific antibodies as assessed by blood test | 3 and 12 months
  Change in positivity of donor specific antibodies from baseline
Change in mean fluorescence index of donor specific antibodies as assessed by blood test | 3 and 12 months
  Change in mean fluorescence index of donor specific antibodies from baseline
Incidence rate of adverse event as assessed by questionnaire | 4 years
  Summary tables of incidence rates for adverse event reporting of participants receiving rituximab in addition to standard of care compared to participants receiving standard of care alone
Health-related quality of life (QoL) as assessed by EuroQoL EQ-5D-5L/EQ-5D-Y questionnaire | 3 months, 1, 2, 3 and 4 years
  A QoL score is obtained according to the answers to the EQ-5D-5L/EQ-5D-Y questionnaires. The QoL score comprises of 2 numbers. The first is a 5-digit number for the EQ-5D-5L descriptive system describing the 5 dimensions asked in the questionnaire. For example 11111 indicates no problems on any of the 5 dimensions whilst 55555 indicates extreme problems on all of the 5 dimensions. The second number is the EQ-VAS (EuroQoL-Visual Analogue Scale) score. This is a value between 0 and 100 where 0 is the worst health the respondent can imagine and 100 is the best health.
Cost effectiveness economic analysis | 4 years
  Statistical decision model built for economic analysis of cost per quality-adjusted life year gained from perspective of the National Health Service

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Willicombe, MA MRCP MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No